CLINICAL TRIAL: NCT03661346
Title: Blood Loss and Visibility With Esmolol vs. Labetalol in Endoscopic Sinus Surgery: A Randomized Trial
Brief Title: Esmolol vs. Labetalol in Endoscopic Sinus Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-0309
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2017-03

CONDITIONS: Chronic Sinusitis
MeSH Terms: interventions — Labetalol; esmolol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esmolol (Experimental): Patients receiving esmolol when intra-operative MAP > 80 mmHg.
  Interventions: Drug: Esmolol
- Labetalol (Active Comparator): Patients receiving labetalol when intra-operative MAP > 80 mmHg
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Labetalol — Aliquots of 20mg of Labetol
  • Maximum Dose - 300mg total for case
  Arms: Labetalol
Drug: Esmolol — Infusion - 0.1mg/kg/min
  • Maximum Dose - after 30 minutes, 0.3mg/kg/min
  Arms: Esmolol

SUMMARY:
The purpose of this study is to compare esmolol and labetalol bleeding and intra-operative visibility scores in functional endoscopic sinus surgery.

DETAILED DESCRIPTION:
BACKGROUND: Improved intraoperative visibility during functional endoscopic sinus surgery (FESS) decreases the risk of serious orbital or skull base injuries. Beta blockers are among several methods used to reduce mean arterial pressure (MAP), heart rate (HR) and mucosal bleeding. Labetalol (mixed alpha-1-beta blocker) reduces HR and MAP; however, its alpha-1 blockade may mitigate topical epinephrine decongestant effects. Esmolol (selective beta-1 blocker) does not have direct antagonistic effects on topical epinephrine. This study compares the hemodynamic parameters (rate of blood loss, MAP control, HR) and intraoperative visibility during FESS between esmolol and labetalol.

ELIGIBILITY:
Inclusion Criteria:

* History of CRS with or without nasal polyps
* Undergoing FESS for CRS
* American Society of Anesthesiologists (ASA) physical status 1 (healthy) or 2 (patient with mild systemic disease).

Exclusion Criteria:

* Pregnancy
* Asthma
* COPD
* Bradycardia
* Heart failure
* End stage renal disease
* Cerebrovascular accident
* Diabetes mellitus
* Preoperative use of NSAIDs, aspirin, or beta-blockers
* Body mass index (BMI) greater than 40 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Chaaban, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months to 3 years at time of publication (if applicable)

RESULTS

PARTICIPANT FLOW:
Groups:
- Esmolol: Patients receiving esmolol when intra-operative MAP > 80 mmHg.
  Esmolol: Infusion - 0.1mg/kg/min
  • Maximum Dose - after 30 minutes, 0.3mg/kg/min
- Labetalol: Patients receiving labetalol when intra-operative MAP > 80 mmHg
  Labetalol: Aliquots of 20mg of Labetol
  • Maximum Dose - 300mg total for case
Period: Overall Study
Arm/Group | Esmolol | Labetalol
Started | 13 (Esmolol administration) | 15
Completed | 13 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with chronic rhinosinusitis undergoing FESS
Groups:
- Total: Total of all reporting groups
Arm/Group | Esmolol | Labetalol | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (17) | 51 (16) | 50 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 10 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Intra-operative Surgical Visibility - Boezaart Scale
Description: Standardized scoring systems used by surgeons to rate surgical field quality in FESS:
  Boezaart scale (0-5):
  0 = no bleeding (optimal)
  1. = slight bleeding with no suction required
  2. = slight bleeding with occasional suctioning required
  3. = slight bleeding with frequent suctioning required
  4. = moderate bleeding with frequent suctioning required and surgical field visibility is compromised when suctioning is removed
  5. = severe bleeding (worst) with constant suctioning required and compromised view
Time Frame: Duration of operation
Population: Those analyzed had complete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmolol | Labetalol
Number analyzed (Participants) | 13 | 15
score on a scale | 3.1 (.69) | 3.1 (.89)

2. Primary Outcome: Intra-operative Surgical Visibility - Wormald Scale
Description: Standardized scoring systems used by surgeons to rate surgical field quality in FESS:
  Wormald scale (0-10):
  0 = No bleeding (optimal)
  1. = 1-2 points of blood ooze
  2. = 3-4 points of ooze
  3. = 5-6 points of ooze
  4. = 7-8 points of ooze
  5. = 9-10 points of ooze
  6. = >10 points of ooze, obscuring field
  7. = Mild field bleeding with slow post-nasal accumulation
  8. = Moderate field bleeding with moderate post-nasal accumulation
  9. = Moderate-severe field bleeding with rapid post-nasal accumulation
  10. = Severe bleeding (worst) with nose filling rapidly
Time Frame: Duration of operation up to 3 hours
Population: Those included had complete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esmolol | Labetalol
Number analyzed (Participants) | 13 | 15
score on a scale | 6.1 (1.7) | 5.9 (1.9)

3. Secondary Outcome: Rate of Blood Loss
Description: milliliters per minute
Time Frame: Duration of operation up to 3 hours
Population: Those included had complete data
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Esmolol | Labetalol
Number analyzed (Participants) | 13 | 15
mL/min | .59 (.28) | .66 (.37)

4. Secondary Outcome: Average Mean Arterial Blood Pressure
Description: units of mmHg, measured throughout operation
Time Frame: Duration of operation up 3 hours/completion of operation
Population: Those included had complete data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Esmolol | Labetalol
Number analyzed (Participants) | 13 | 15
mmHg | 79.7 (7.5) | 79.4 (7.7)

5. Secondary Outcome: Average Heart Rate
Description: units of beats per minute, measured throughout the operation
Time Frame: Duration of operation up to 3 hours/completion of surgery
Population: Those included had complete data
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Esmolol | Labetalol
Number analyzed (Participants) | 13 | 15
bpm | 72 (8.7) | 69 (11.7)

ADVERSE EVENTS:
Time Frame: Adverse events collected following surgery in recovery room
Arm/Group | Esmolol | Labetalol
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03661346/SAP_001.pdf
  • Study Protocol (2016-01-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT03661346/Prot_003.pdf
  • Informed Consent Form (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT03661346/ICF_004.pdf